CLINICAL TRIAL: NCT05348239
Title: A Phase II Study to Evaluate Oral Chlorophyllin in Hemorrhagic Cystitis Secondary to Radiation Therapy for Pelvic Malignancies
Brief Title: Chlorophyllin Tablets for Urinary Bleeding Following Radiation Therapy for Cancers of Pelvic Organs
Acronym: CLARITY
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tata Memorial Centre (Other)
Collaborators: Bhabha Atomic Research Centre (BARC), Mumbai (Unknown)
Responsible Party: Principal Investigator, Dr Gagan Prakash, Professor, Urologic Oncology, Tata Memorial Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 900878
Record Dates: First submitted 2022-03-17; First posted 2022-04-27 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Hemorrhagic Cystitis
MeSH Terms: conditions — Cystitis, Hemorrhagic | interventions — chlorophyllin

STUDY DESIGN:
Intervention Model Description: A prospective, single centre, single-arm, interventional phase II study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oral Chlorophyllin arm (Experimental): Participants will receive oral Sodium Copper Chlorophyllin at a dose of 750mg once daily (OD) on an empty stomach.
  Interventions: Drug: Sodium Copper Chlorophyllin

INTERVENTIONS:
Drug: Sodium Copper Chlorophyllin — Sodium-copper-chlorophyllin (CHL) is a phytopharmaceutical drug obtained from green plant pigment, chlorophyll. Chlorophyllin scavenges radiation-induced free radicals and reactive oxygen species. It is used as a food colorant and OTC in the USA, Japan, Australia and China for many years for a variety of health benefits including prevention of body odour in geriatric patients, enhanced wound healing, antibacterial action, prevention of cancer in the high-risk populations exposed to hepatocarcinogen aflatoxin B1, treatment of faecal incontinence etc. Studies have shown that CHL has immunostimulatory, anti-inflammatory and antiviral effects in addition to antioxidant and radioprotective properties. It increases the expression of a transcription factor (protein) Nrf2 which improves lymphocyte survival and enables efficient detoxification after exposure to radiation. The duration of therapy will be up to 6 months depending upon the response of participants.

SUMMARY:
To assess the efficacy of oral chlorophyllin tablets for urinary bleeding following radiation therapy for cancers of pelvic organs.

DETAILED DESCRIPTION:
Radiation therapy to the pelvis is a commonly used treatment modality for urological, gynaecological and rectal cancers. Intensity modulation and image guidance have improved the delivery of radiation therapy in recent times. However, this does not eliminate the risk of radiation-induced damage to the adjacent healthy tissue - in this consideration, the bladder. Hemorrhagic cystitis accounts for 5-7% of emergency urology admissions. The procedure for the management of radiation cystitis proceeds from non-invasive oral drugs and HBOT to minimally invasive treatment like intravesical therapy and angioembolization, to more morbid procedures like cystectomy and urinary diversion. Although these treatment modalities have shown some success, most patients continue to have recurrent/persistent hematuria. There is a need to explore options of other oral/intravesical agents which can aid in mucosal healing and stop hematuria with lasting effects. Sodium-copper-chlorophyllin (CHL) is a phytopharmaceutical drug obtained from green plant pigment, chlorophyll. It is a semi-synthetic mixture of sodium copper salts derived from chlorophyll. Chlorophyllin scavenges radiation-induced free radicals and reactive oxygen species. Research at BARC has shown that chlorophyllin prevents radiation-induced toxicity in normal hematopoietic tissues and normal epithelial cells. A phase 1 clinical study in healthy volunteers indicate that CHL is safe and tolerable in humans and has not shown any severe adverse events. The purpose of this study is to evaluate the safety and efficacy of oral sodium copper chlorophyllin in hemorrhagic cystitis secondary to radiation therapy for pelvic malignancy.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age with a history of radiotherapy for pelvic malignancy in the past more than 3 months back.
* Any grade of radiation-induced cystitis as per RTOG criteria (RTOG Grade 1-4 equivalent to CTCAE Grade 1-3).
* Adequate liver function defined as ALT/ALT ≤ 3 times ULN and total bilirubin ≤ 2 times ULN. Elevated transaminases up to 5 times ULN is allowed in patients with liver metastasis.
* Adequate renal function defined as creatine clearance ≥ 30 mL/min (By Cockcroft-Gault formula).

Exclusion Criteria:

* Known hypersensitivity or contraindications against sodium chlorophyllin.
* Hemodynamically unstable patients not responding to initial resuscitation.
* Patients with life-threatening hemorrhagic cystitis requiring urgent invasive intervention (CTCAE grade 4).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-03-26 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of Objective Response Rate (ORR) as per CTCAE v5.0. | Baseline
  Objective Response Rate (ORR) The proportion of patients with CR/PR.The ORR will be determined as below.Complete response(CR):resolution of hematuria (gross/macroscopic hematuria for grade II/III and microscopic hematuria for grade I hemorrhagic cystitis) Partial response(PR):improvement (decrease by at least 1 grade of hemorrhagic cystitis but not complete resolution of hematuria over 3 months from the start of treatment.The grading of hemorrhagic cystitis will be as per the CTCAE v5.0.
Assessment of Objective Response Rate (ORR) as per CTCAE v5.0. | Post 1 month
  Objective Response Rate (ORR) The proportion of patients with CR/PR.The ORR will be determined as below.Complete response(CR):resolution of hematuria (gross/macroscopic hematuria for grade II/III and microscopic hematuria for grade I hemorrhagic cystitis) Partial response(PR):improvement (decrease by at least 1 grade of hemorrhagic cystitis but not complete resolution of hematuria over 3 months from the start of treatment.The grading of hemorrhagic cystitis will be as per the CTCAE v5.0.
Assessment of Objective Response Rate (ORR) as per CTCAE v5.0. | Post 3 months
  Objective Response Rate (ORR) The proportion of patients with CR/PR.The ORR will be determined as below.Complete response(CR):resolution of hematuria (gross/macroscopic hematuria for grade II/III and microscopic hematuria for grade I hemorrhagic cystitis) Partial response(PR):improvement (decrease by at least 1 grade of hemorrhagic cystitis but not complete resolution of hematuria over 3 months from the start of treatment.The grading of hemorrhagic cystitis will be as per the CTCAE v5.0.
Assessment of Objective Response Rate (ORR) as per CTCAE v5.0. | Post 6 months
  Objective Response Rate (ORR) The proportion of patients with CR/PR.The ORR will be determined as below.Complete response(CR):resolution of hematuria (gross/macroscopic hematuria for grade II/III and microscopic hematuria for grade I hemorrhagic cystitis) Partial response(PR):improvement (decrease by at least 1 grade of hemorrhagic cystitis but not complete resolution of hematuria over 3 months from the start of treatment.The grading of hemorrhagic cystitis will be as per the CTCAE v5.0.

SECONDARY OUTCOMES:
Assessment of Bladder Cancer Index (BCI) scores. | Baseline, post 1 month, post 3 months
  Bladder cancer index (BCI) scores will be calculated at baseline, 1 month and 3 months for each study participant.
  Minimum value - 0, Maximum value - 100, Higher scores depict better outcome.
Assessment of Treatment Failure (TF). | Post 3 months
  Treatment Failure (TF) defined as requirement of alternative intervention for persistent severe hematuria within 3 months from the start of treatment or early stoppage due to intolerable side effects in the absence of PR/CR [Intervention: multiple cystoscopies with clot evacuation, cystectomy, hyperbaric oxygen therapy (HBOT) or transfusion due to persistent drop in hemoglobin].
Evaluation of treatment failure-free survival. | Baseline to up to 3 months
  Treatment failure-free survival is defined as the time from enrolment to the date of first intervention up to 3 months or date of discontinuation of therapy due to intolerable side effects in the absence of PR/CR.
Assessment of Quality of Life (QOL) using EORTC -QLQ C-30 questionnaire. | Baseline, post 1 month, post 3 months
  QoL will be measured using the EORTC-QLQ-30 questionnaire at baseline, 1 month and 3 months for each study participant.
  Minimum value - 0, Maximum value cannot be predetermined. five functional scales (physical, role, cognitive, emotional, and social), three symptom scales (fatigue, pain, and nausea and vomiting), a global health status / QoL scale, and a number of single items assessing additional symptoms commonly reported by cancer patients (dyspnoea, loss of appetite, insomnia, constipation and diarrhoea) and perceived financial impact of the disease. Therefore, higher scores depict better outcomes for some scales whereas for some scales lower scores depict better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Gagan Prakash, Principal Investigator — Tata Memorial Centre
Locations (1):
- Tata Memorial Centre, Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No
All study-related information will be strictly maintained and will be shared only with the IEC and DSMB authorities.

REFERENCES:
- [Background] Smit SG, Heyns CF. Management of radiation cystitis. Nat Rev Urol. 2010 Apr;7(4):206-14. doi: 10.1038/nrurol.2010.23. Epub 2010 Mar 9. PMID 20212517
- [Background] Browne C, Davis NF, Mac Craith E, Lennon GM, Mulvin DW, Quinlan DM, Mc Vey GP, Galvin DJ. A Narrative Review on the Pathophysiology and Management for Radiation Cystitis. Adv Urol. 2015;2015:346812. doi: 10.1155/2015/346812. Epub 2015 Dec 22. PMID 26798335
- [Background] Sandhu SS, Goldstraw M, Woodhouse CR. The management of haemorrhagic cystitis with sodium pentosan polysulphate. BJU Int. 2004 Oct;94(6):845-7. doi: 10.1111/j.1464-410X.2004.05044.x. PMID 15476520
- [Background] Feldmeier JJ, Hampson NB. A systematic review of the literature reporting the application of hyperbaric oxygen prevention and treatment of delayed radiation injuries: an evidence based approach. Undersea Hyperb Med. 2002 Spring;29(1):4-30. PMID 12507182
- [Background] Oscarsson N, Muller B, Rosen A, Lodding P, Molne J, Giglio D, Hjelle KM, Vaagbo G, Hyldegaard O, Vangedal M, Salling L, Kjellberg A, Lind F, Ettala O, Arola O, Seeman-Lodding H. Radiation-induced cystitis treated with hyperbaric oxygen therapy (RICH-ART): a randomised, controlled, phase 2-3 trial. Lancet Oncol. 2019 Nov;20(11):1602-1614. doi: 10.1016/S1470-2045(19)30494-2. Epub 2019 Sep 16. PMID 31537473
- [Background] Villeirs L, Tailly T, Ost P, Waterloos M, Decaestecker K, Fonteyne V, Van Praet C, Lumen N. Hyperbaric oxygen therapy for radiation cystitis after pelvic radiotherapy: Systematic review of the recent literature. Int J Urol. 2020 Feb;27(2):98-107. doi: 10.1111/iju.14130. Epub 2019 Oct 15. PMID 31617263
- [Background] Lojanapiwat B, Sripralakrit S, Soonthornphan S, Wudhikarn S. Intravesicle formalin instillation with a modified technique for controlling haemorrhage secondary to radiation cystitis. Asian J Surg. 2002 Jul;25(3):232-5. doi: 10.1016/S1015-9584(09)60181-0. PMID 12376221
- [Background] Westerman ME, Boorjian SA, Linder BJ. Safety and efficacy of intravesical alum for intractable hemorrhagic cystitis: A contemporary evaluation. Int Braz J Urol. 2016 Nov-Dec;42(6):1144-1149. doi: 10.1590/S1677-5538.IBJU.2015.0588. PMID 27509371
- [Background] Comploj E, Pycha A, Trenti E, Palermo S, Bonatti M, Krause P, Folchini DM, Pycha A. Transarterial Embolization in the Management of Intractable Haemorrhage. Urol Int. 2021;105(1-2):95-99. doi: 10.1159/000511123. Epub 2020 Oct 16. PMID 33070141
- [Background] Linder BJ, Tarrell RF, Boorjian SA. Cystectomy for refractory hemorrhagic cystitis: contemporary etiology, presentation and outcomes. J Urol. 2014 Dec;192(6):1687-92. doi: 10.1016/j.juro.2014.06.030. Epub 2014 Jun 14. PMID 24936722
- [Background] Chlorophyll and Chlorophyllin Linus Pauling Institute Oregon State University. (Micronutrient Information)
- [Background] Egner PA, Wang JB, Zhu YR, Zhang BC, Wu Y, Zhang QN, Qian GS, Kuang SY, Gange SJ, Jacobson LP, Helzlsouer KJ, Bailey GS, Groopman JD, Kensler TW. Chlorophyllin intervention reduces aflatoxin-DNA adducts in individuals at high risk for liver cancer. Proc Natl Acad Sci U S A. 2001 Dec 4;98(25):14601-6. doi: 10.1073/pnas.251536898. Epub 2001 Nov 27. PMID 11724948
- [Background] Citrin D, Cotrim AP, Hyodo F, Baum BJ, Krishna MC, Mitchell JB. Radioprotectors and mitigators of radiation-induced normal tissue injury. Oncologist. 2010;15(4):360-71. doi: 10.1634/theoncologist.2009-S104. PMID 20413641
- [Background] Oriya A, Takahashi K, Inanami O, Miura T, Abe Y, Kuwabara M, Kashiwakura I. Individual differences in the radiosensitivity of hematopoietic progenitor cells detected in steady-state human peripheral blood. J Radiat Res. 2008 Mar;49(2):113-21. doi: 10.1269/jrr.07079. Epub 2007 Dec 12. PMID 18075225
- [Background] Dainiak N. Hematologic consequences of exposure to ionizing radiation. Exp Hematol. 2002 Jun;30(6):513-28. doi: 10.1016/s0301-472x(02)00802-0. PMID 12063018
- [Background] Jubert C, Mata J, Bench G, Dashwood R, Pereira C, Tracewell W, Turteltaub K, Williams D, Bailey G. Effects of chlorophyll and chlorophyllin on low-dose aflatoxin B(1) pharmacokinetics in human volunteers. Cancer Prev Res (Phila). 2009 Dec;2(12):1015-22. doi: 10.1158/1940-6207.CAPR-09-0099. Epub 2009 Dec 1. PMID 19952359
- [Background] Nagini S, Palitti F, Natarajan AT. Chemopreventive potential of chlorophyllin: a review of the mechanisms of action and molecular targets. Nutr Cancer. 2015;67(2):203-11. doi: 10.1080/01635581.2015.990573. Epub 2015 Feb 4. PMID 25650669
- [Background] Nahata MC, Slencsak CA, Kamp J. Effect of chlorophyllin on urinary odor in incontinent geriatric patients. Drug Intell Clin Pharm. 1983 Oct;17(10):732-4. doi: 10.1177/106002808301701006. PMID 6628224
- [Background] Christiansen SB, Byel SR, Stromsted H, Stenderup JK, Eickhoff JH. [Can chlorophyll reduce fecal odor in colostomy patients?]. Ugeskr Laeger. 1989 Jul 3;151(27):1753-4. Danish. PMID 2675439
- [Background] Yamazaki H, Fujieda M, Togashi M, Saito T, Preti G, Cashman JR, Kamataki T. Effects of the dietary supplements, activated charcoal and copper chlorophyllin, on urinary excretion of trimethylamine in Japanese trimethylaminuria patients. Life Sci. 2004 Apr 16;74(22):2739-47. doi: 10.1016/j.lfs.2003.10.022. PMID 15043988
- [Background] WEINGARTEN M, PAYSON B. Deodorization of colostomies with chlorophyll. Rev Gastroenterol. 1951 Aug;18(8):602-4. No abstract available. PMID 14864969
- [Background] BOWERS WF. Chlorophyll in wound healing and suppurative disease. Am J Surg. 1947 Jan;73(1):37-50. doi: 10.1016/0002-9610(47)90287-0. No abstract available. PMID 20279378
- [Background] CARPENTER EB. Clinical experiences with chlorophyll preparations with particular reference to chronic osteomyelitis and chronic ulcers. Am J Surg. 1949 Feb;77(2):167-71. doi: 10.1016/0002-9610(49)90419-5. No abstract available. PMID 18108595
- [Background] 2004 Physicians' Desk Reference. 58th ed. Stamford: Thomson Health Care, Inc.; 2003.
- [Background] Smith RG. Enzymatic debriding agents: an evaluation of the medical literature. Ostomy Wound Manage. 2008 Aug;54(8):16-34. PMID 18716339
- [Background] Weir D, Farley KL. Relative delivery efficiency and convenience of spray and ointment formulations of papain/urea/chlorophyllin enzymatic wound therapies. J Wound Ostomy Continence Nurs. 2006 Sep-Oct;33(5):482-90. doi: 10.1097/00152192-200609000-00005. PMID 17133135
- [Background] Aggarwal A, Shrivastava A, Kumar A, Ali A. Clinical and Epidemiological Features of SARS-CoV-2 Patients in SARI Ward of a Tertiary Care Centre in New Delhi. J Assoc Physicians India. 2020 Jul;68(7):19-26. PMID 32602676
- [Background] Suryavanshi S, Sharma D, Checker R, Thoh M, Gota V, Sandur SK, Sainis KB. Amelioration of radiation-induced hematopoietic syndrome by an antioxidant chlorophyllin through increased stem cell activity and modulation of hematopoiesis. Free Radic Biol Med. 2015 Aug;85:56-70. doi: 10.1016/j.freeradbiomed.2015.04.007. Epub 2015 Apr 11. PMID 25872101
- [Background] Sharma D, Kumar SS, Sainis KB. Antiapoptotic and immunomodulatory effects of chlorophyllin. Mol Immunol. 2007 Jan;44(4):347-59. doi: 10.1016/j.molimm.2006.02.031. Epub 2006 Apr 17. PMID 16616780
- [Background] Warny M, Helby J, Nordestgaard BG, Birgens H, Bojesen SE. Lymphopenia and risk of infection and infection-related death in 98,344 individuals from a prospective Danish population-based study. PLoS Med. 2018 Nov 1;15(11):e1002685. doi: 10.1371/journal.pmed.1002685. eCollection 2018 Nov. PMID 30383787
- [Background] Tan L, Wang Q, Zhang D, Ding J, Huang Q, Tang YQ, Wang Q, Miao H. Lymphopenia predicts disease severity of COVID-19: a descriptive and predictive study. Signal Transduct Target Ther. 2020 Mar 27;5(1):33. doi: 10.1038/s41392-020-0148-4. No abstract available. PMID 32296069
- [Background] Zhang X, Tan Y, Ling Y, Lu G, Liu F, Yi Z, Jia X, Wu M, Shi B, Xu S, Chen J, Wang W, Chen B, Jiang L, Yu S, Lu J, Wang J, Xu M, Yuan Z, Zhang Q, Zhang X, Zhao G, Wang S, Chen S, Lu H. Viral and host factors related to the clinical outcome of COVID-19. Nature. 2020 Jul;583(7816):437-440. doi: 10.1038/s41586-020-2355-0. Epub 2020 May 20. PMID 32434211
- [Background] Ye Q, Wang B, Mao J. The pathogenesis and treatment of the ;Cytokine Storm' in COVID-19. J Infect. 2020 Jun;80(6):607-613. doi: 10.1016/j.jinf.2020.03.037. Epub 2020 Apr 10. PMID 32283152
- [Background] Interim Clinical Study Report (Project No. 0462-16) - An Open Label, Clinical Study To Assess Safety, Tolerability, Pharmacokinetics And Pharmacodynamics Of Sodium Copper Chlorophyllin In Healthy Adult, Human Male Subjects.